CLINICAL TRIAL: NCT06899776
Title: Assessing Chest Pain Using Point-of-Care High-Sensitivity Troponin I in the Emergency Department
Acronym: ACUTE
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Abbott Point of Care (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00117677
Record Dates: First submitted 2025-03-05; First posted 2025-03-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: ACS (Acute Coronary Syndrome)
Keywords: chest pain; myocardial infarction; Emergency Department
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Myocardial Infarction; Emergencies | interventions — Surgical Instruments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with possible ACS: Adult Emergency Department patients with symptoms suggestive of acute coronary syndrome undergoing a standard-of-care evaluation possible acute coronary syndrome (ACS) in the ED including blood testing for hs-cTnI (Beckman Coulter) completed in a core laboratory.
  Interventions: Device: Abbott i-STAT point of care (POC) device

INTERVENTIONS:
Device: Abbott i-STAT point of care (POC) device — During the study period all ED patients with chest pain will have an extra lithium heparin blood sample obtained for each troponin test ordered and collected in the ED (typically 2, but this may range from 1-3 troponin measures), which will be used for immediate hs-cTnI measurement by research personnel using an Abbott i-STAT POC device.

SUMMARY:
The goal of this proposal is to improve the quality and value of care for patients with acute chest pain by investigating the potential impact of point-of-care (POC) high sensitivity cardiac troponin (hs-cTn) testing in the Emergency Department (ED) and exploring how best to integrate POC hs-cTnl into ED risk stratification workflows. The study hypothesizes that the Abbott i-STAT POC hs-cTnI assay will decrease time-to-result (TTR) and ED length of stay (LOS), while increasing ED revenue for patients with acute chest pain compared to a strategy of central laboratory hs-cTnI testing.

DETAILED DESCRIPTION:
Use of point-of-care (POC) testing in the Emergency Department (ED) has been previously established as a method to reduce the time-to-disposition-decision (TTD) making for emergency physicians, which in-turn can reduce ED length of stay (LOS) and time-to-treatment (TTT) of time sensitive conditions, such as myocardial infarctions (MIs). Recently, new POC high sensitivity cardiac troponin I (hs-cTnI) assays have been developed which offer similar diagnostic performance to traditional central lab hs-cTnI testing. However, data examining POC hs-cTnI measurement in U.S. ED settings are limited. In particular, studies have yet to evaluate the potential impact of POC hs-cTnI implementation on time to troponin result (TTR), time-to-last-troponin-result (TTLT), time-to-disposition-decision (TTD), time-to-treatment (TTT), and ED LOS. In addition, limited data exists on how best to implement POC hs-cTnI into ED clinical practice, such as whether POC hs-cTnI measures should be paired with a risk score or incorporated into an accelerated diagnostic protocol.

This record is a prospective multisite observational cohort study of 600 adult ED patients with symptoms suggestive of acute coronary syndrome and without ST-segment elevation myocardial infarction (STEMI) across 3 EDs. Participants, accrued under a waiver of informed consent, will undergo a standard-of-care evaluation for possible acute coronary syndrome (ACS) in the ED including blood testing for hs-cTnI (Beckman Coulter) completed in a central laboratory. During the study period all ED patients with chest pain will have an extra lithium heparin blood sample obtained for each troponin test ordered and collected in the ED (typically 2, but this may range from 1-3 troponin measures), which will be used for immediate hs-cTnI measurement by research personnel using an Abbott i-STAT Alinity. Clinicians will be blinded to the POC hs-cTnI results and will base clinical decisions on central laboratory hs-cTn measures. Blood draw times, result times for point-of-care (POC) and central laboratory measures, patient ED arrival, patient ED bedded, ED disposition decision times, and ED discharge times will be recorded on all patients. Following each POC hs-cTnI measurement the treating attending physician will be surveyed regarding whether a negative or positive POC result would change ED disposition or treatment including time stamps to determine estimated TTD, ED LOS and TTT for the POC hs-cTnI measurement strategy. Data from these surveys will be compared to actual TTD, ED LOS and treatment times based on the central laboratory hs-cTnI measurement strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to18 years
* Symptoms suggestive of acute coronary syndrome:
* Acute chest, epigastric, neck, jaw or arm pain or discomfort or pressure without apparent non-cardiac source
* Shortness of breath, nausea, vomiting, fatigue/malaise, or
* Other equivalent discomfort suggestive of an myocardial infarction (MI)
* Electrocardiogram (ECG) ordered as part of standard of care
* At least one troponin collected as standard of care
* Study specific blood sample collected within ± 5 minutes of clinical draw

Exclusion Criteria:

* ST-segment elevation myocardial infarction (STEMI) Activation
* Unstable vitals signs: symptomatic hypotension at the time of enrollment (systolic < 90 mm Hg), tachycardia (HR>120), bradycardia (HR<40), and hypoxemia (<90% pulse-oximetry on room air or normal home oxygen flow rate)
* Central laboratory hs-cTn testing resulted or in process (>5 minutes) prior to study accrual
* Prior enrollment
* Terminal diagnosis with life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years old) presenting to the ED with symptoms concerning for acute coronary syndrome (ACS) and an ECG and troponin ordered as part of standard of care, will be eligible for accrual. Patients with STEMI activation or unstable vital signs will be excluded. In addition, patients will be required to have a (extra) lithium heparin blood sample collected within ± 5 minutes of their clinical draw for hs-cTnI. Patients with central laboratory hs-cTnI testing or a hs-cTnI measure resulted prior to study accrual also be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time-to-result (TTR) of hs-cTnI | Index visit to Hour 24
  Defined as the time from blood collection to result time of the hs-cTnI assay, as recorded by research staff for the Abbott i-STAT POC device and by the electronic health record for central lab Beckman Coulter Access 2 hs-cTnI measures. TTR will be collected for each troponin test ordered and collected in the Emergency Department (typically two tests per patient).

SECONDARY OUTCOMES:
Time-to-last-troponin-result (TTLT) | Index visit to Hour 24
  Defined as the time from ED arrival to the result time of the last hs-cTnI measure in the ED (by the POC and central lab strategies).
Time-to-disposition decision (TTD) | Index visit to Hour 24
  Defined as the time from the patient being bedded in the ED to provider decision on disposition (discharge vs admission).
ED length of stay (LOS) | Index visit to Hour 72
  Defined as the time from ED arrival to disposition (discharged, admitted, observation unit, left against medical advice, transfer, etc.).
ED Revenue amount | Index visit to Month 6
  Calculate the associated ED revenue generated based on an average of $550 in revenue per bed-hour.
Time-to-treatment (TTT) | Index visit to Hour 24
  Defined by the time from the patient being bedded in the ED to the provider's decision to initiate treatment for patients with a Type 1 Non-ST-Segment Elevation Myocardial Infarction (NSTEMI) diagnosis (e.g., heparin drip).
Number of Myocardial Infarctions (MI) | Baseline and Week 1
  Number of Myocardial Infarctions (MI)
Number of Cardiac Deaths | Baseline and Day 30
  Number of Cardiac Deaths

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mahler, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Carolinas Medical Center, Charlotte, North Carolina
  - High Point Medical Center, High Point, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT06899776/Prot_SAP_000.pdf